CLINICAL TRIAL: NCT01346319
Title: A Randomized Double-Blind, Placebo-controlled Dose Escalating Study of the Pharmacokinetics, Safety and Tolerability of Testosterone Undecanoate (ABT-SLV361) in Hypogonadal Males
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of Testosterone Undecanoate in Hypogonadal Males.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M12-778
Record Dates: First submitted 2011-04-20; First posted 2011-05-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-09

CONDITIONS: Hypogonadal Males
Keywords: dose escalating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone undecanoate (Active Comparator)
  Interventions: Drug: ABT-SLV361
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-SLV361 — For dose groups 1, 2 and 3 medication is taken 1 time per day the first day followed by 2 times per day for 14 days. For dose groups 4 and 5, medication is taken 1 time per day for the first day followed by 2 times per day for 28 days.
  Arms: Testosterone undecanoate
Drug: placebo — For dose groups 1, 2 and 3 medication is taken 1 time per day the first day followed by 2 times per day for 14 days. For dose groups 4 and 5, medication is taken 1 time per day for the first day followed by 2 times per day for 28 days.
  Arms: Placebo

SUMMARY:
Phase 1 Dose Escalating Study of the safety, tolerability and pharmacokinetics of testosterone in hypogonadal males.

DETAILED DESCRIPTION:
M12-778 is a rising multiple dose, randomized, double blind, placebo controlled single center study. It will have 5 dose groups of 20 subjects in dose groups 1,2 and 3 and 24 subjects in dose groups 4 and 5; a total of 84 subjects . There will be a 7 day period between dose groups 1,2 and 3 to assess the safety of increasing to the next dose. Dose groups of 4 and 5 will be run in parallel. Subjects will be confined in center for 20 days for dose groups 1,2 and 3 and 33 days for dose groups 4 and 5.

ELIGIBILITY:
Inclusion Criteria

1. Serum total testosterone < 300 ng/dL based on two blood samples obtained between 6 and 10 AM on two separate occasions at least 48 hours apart. Previously documented total testosterone results obtained within 6 weeks of Study Day -2 may be used during screening for subjects not currently on androgen replacement therapy, or following washout of androgen replacement therapy.
2. Subjects naïve to androgen replacement or washout of 12 weeks following intramuscular androgen injections; 4 weeks following topical or buccal androgens; and 3 weeks following oral androgens. Washout should be completed by Study Day -2.
3. Subject is judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12 lead electrocardiogram (ECG) performed at Screening.
4. Must voluntarily sign and date each informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria

1. History of significant sensitivity or allergy to any drug, including androgens, castor oil or product excipients.
2. Previous history or current or suspected prostate or breast cancer, and/or previous history of cancer (except basal cell carcinoma of the skin).
3. Subjects not on a stable medication regimen for at least three months for the treatment of a chronic condition such as hypertension, hyperlipidemia or diabetes mellitus.
4. Use of known inhibitors (e.g., ketoconazole) or inducers (e.g., dexamethasone, phenytoin, rifampin, carbamazepine) of cytochrome P450 3A (CYP3A) within 30 days prior to study drug administration and through the end of the study.
5. Use of any drug within 5 half-lives of the last dose in the past 6 months prior to Study Day -2 without principal investigator and/or sponsor approval.
6. Receipt of any drug by injection within 30 days or 10 half-lives (which ever is longer) prior to study drug administration without principal investigator and/or sponsor approval.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetics of testosterone after multiple oral doses of ABT-SLV361 in hypogonadal males | During confinement
  Blood sample results for testosterone

SECONDARY OUTCOMES:
To determine the pharmacokinetic of testosterone undecanoate after multiple oral doses of ABT-SLV361 in hypogonadal males | During confinement
  Blood sample results for testosterone undecanoate

CONTACTS AND LOCATIONS:
Overall Officials: Bela Denes, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 51964, Fort Myers, Florida, United States